CLINICAL TRIAL: NCT01492946
Title: Impaired Preoperative Nutritional Status as a Risk Factor for Postoperative Clinical Outcome (PreopBIA)
Brief Title: Impaired Preoperative Nutritional Status as a Risk Factor for Postoperative Clinical Outcome
Acronym: PreopBIA
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia Spies, study director, Charite University, Berlin, Germany
Other Study IDs: PreopBIA
Record Dates: First submitted 2011-12-14; First posted 2011-12-15 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Nutritional Status
Keywords: Malnutrition; Post-operative outcome; Phase angle; MUST; Clavien Dindo classification; Bioelectrical impedance analysis
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Elective surgical patients: Elective surgical patients in the Charité University Berlin Campus Charité Mitte

SUMMARY:
The aim of this retrospective observational study is to determine the impact of preoperative nutritional status on postoperative outcome. Elective surgical patients were screened with Bio-Impedance-Analysis, Malnutritional Universal Screening Tool, and other variables for body composition. Outcome parameters were collected by patient chart review.

ELIGIBILITY:
Inclusion Criteria:

1. Elective surgical intervention
2. Patients must be 18 years or older
3. Ambulation
4. ASA-Score I-IV
5. bioelectrical impedance analysis to determine the phase angle

Exclusion Criteria:

1. Emergency surgery
2. Pregnancy
3. ASA Score V-VI
4. Amputated limbs
5. Pacemaker and defibrillators
6. Cerebrovascular events
7. Tattoos on the electrode locations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Elective surgical patients
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2010-05; Primary Completion 2010-11 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Phase-angle | preoperative

SECONDARY OUTCOMES:
body weight | preoperative
body mass index (BMI) | preoperative
preoperative weight loss | 3 month weight loss before operation
hip/waist ratio | preoperative
Malnutrition Universal Screening Tool (MUST) | preoperative
  The MUST is recommended by ESPEN as the preferred screening tool for patients in the community (Kondrup J et al., Clinical Nutrition 2003; 22: 415-421)
postoperative complications | postoperative
  The Clavien-Dindo Classification of Surgical Complications (Dindo D., Demartines N., Clavien P.A.; Ann Surg. 2004; 244: 931-937)
Length of hospital stay | participants will be followed for the duration of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD Prof., Study Director — Department of Anesthesiology and Operative Intensive Care Medicine Campus Charité Mitte, Charite University, Berlin, Germany
Locations (1):
- Department of Anesthesiology and Operative Intensive Care Medicine Campus Charité Mitte, Charite University,, Berlin, State of Berlin, Germany